CLINICAL TRIAL: NCT01735994
Title: Healthy Weight Intervention in Female Athletes: A Randomized Controlled Trial
Brief Title: Efficacy of the Female Athlete Body Project (FAB)
Acronym: FAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tiffany Stewart, Director, Behavior Technology Laboratory, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PBRC 11032; R01MH094448 (NIH)
Record Dates: First submitted 2012-11-14; First posted 2012-11-28 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Eating Disorders; Female Athlete Triad
Keywords: Eating disorders; body image; female athletes; female athlete triad; eating disorder prevention; cluster randomization; risk factors; prevention
MeSH Terms: conditions — Feeding and Eating Disorders; Female Athlete Triad Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Weight Intervention (Experimental): Eating Disorder Prevention Program
  Interventions: Behavioral: Healthy Weight
- Brochure wait list (Other): Brochure wait list control group
  Interventions: Other: Brochure

INTERVENTIONS:
Behavioral: Healthy Weight — Eating Disorder Prevention Program for Athletes
  Arms: Healthy Weight Intervention
Other: Brochure — Brochure on the Female athlete triad
  Arms: Brochure wait list

SUMMARY:
Given the cost of treating eating disorders and the substantial morbidity and mortality associated with these disorders, prevention of eating disorders has considerable public health significance. Female athletes represent an important population for prevention due to their risk for the Female Athlete Triad, which includes inadequate energy intake, irregular or cessation of menses, and osteoporosis. The proposed randomized controlled trial will provide important information regarding the efficacy, acceptability, and feasibility of implementing a brief eating disorder prevention and healthy living program within an existing social system of female athletes.

DETAILED DESCRIPTION:
Research supports the use of a Healthy Weight (HW) program targeting small lifestyle modifications in the prevention of ED onset and in reducing ED risk factors. Studies show that HW can be tailored for specific social systems (e.g., sororities) which can facilitate dissemination and that undergraduate peer-leaders can implement these programs. Interventions that can be administered affordably by endogenous providers are more likely to be disseminated, as indicated by the large scale dissemination of a peer-led ED prevention program by a national sorority. Another target social system for dissemination of ED prevention is collegiate athletics. Research suggests that disordered eating among female athletes is prevalent, and that this group is at greater, or at least equal, risk for developing EDs as non-athlete females. Disordered eating is especially dangerous in female athletes because it increases risk for the Female Athlete Triad (i.e., low energy availability/disordered eating, menstrual disorders, and decreased bone mineral density/osteoporosis) and subsequent injury. Moreover, the triad puts athletes at risk for serious long-term health consequences, such as osteoporosis, reproductive disorders, and cardiovascular disease. Despite this, efforts aimed at prevention of EDs among this group remain surprisingly limited. A pilot study with female athletes suggests that a modified version of HW can be successfully implemented by peer-leaders within the constraints of a competitive athletics program with positive effects at 12 month follow-up. The proposed study is to evaluate a randomized controlled trial of the HW intervention among female athletes. 500 female collegiate athletes from three sites will be randomized to either the HW prevention program or a brochure waitlist control condition using group (cluster) randomization based on teams. Participants will complete surveys and telephone interviews at pretest, posttest, and at 6 and 12 month follow-ups. The investigators will examine; (1) the efficacy of HW in reducing empirically supported ED risk factors relative to a waitlist brochure control condition at one year, (2) whether HW impacts secondary outcomes, including knowledge and identification of the female athlete triad, treatment seeking for the triad, affect, and health care utilization, and (3) whether positive effects for HW replicate the effects from the pilot study at one year and 18 months for the HW condition only. Based on previous promising findings, the department of athletics involved in the study have chosen to implement HW to all athletics teams on a mandatory basis on a staggered schedule. Given that it is unethical to require human subjects to participate in research, the proposed study (i.e., the study) must be separated from the program (i.e., the athlete prevention program) it aims to assess. Thus, the overall study will evaluate (via assessment measures) the program that the departments of athletics deliver at three sites, i.e. LSU, TU/IW, and AU.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Member of a University-sponsored athletic team,
* Are willing and able to provide informed consent, attend all study visits, and comply with the study protocol

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2012-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany M Stewart, PhD, Principal Investigator — Pennington Biomedical
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stewart TM, Pollard T, Hildebrandt T, Beyl R, Wesley N, Kilpela LS, Becker CB. The Female Athlete Body (FAB) study: Rationale, design, and baseline characteristics. Contemp Clin Trials. 2017 Sep;60:63-71. doi: 10.1016/j.cct.2017.06.005. Epub 2017 Jun 10. PMID 28611008
- [Background] Stewart TM, Pollard T, Hildebrandt T, Wesley NY, Kilpela LS, Becker CB. The Female Athlete Body project study: 18-month outcomes in eating disorder symptoms and risk factors. Int J Eat Disord. 2019 Nov;52(11):1291-1300. doi: 10.1002/eat.23145. Epub 2019 Jul 27. PMID 31350934
- [Derived] Stewart T, Kilpela L, Wesley N, Baule K, Becker C. Psychometric properties of the contextual body image questionnaire for athletes: a replication and extension study in female collegiate athletes. J Eat Disord. 2021 May 5;9(1):59. doi: 10.1186/s40337-021-00414-8. PMID 33952348

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment began at the schools in August 2012 and completed in October 2014.
Pre-assignment Details: Only one athlete decided to participate in the prevention program without participating in the study.
Units Other Than Participants: teams
Period: Overall Study
Arm/Group | Healthy Weight Intervention | Brochure Wait List
Started | 263; 13 teams | 218; 15 teams
Post Intervention (3 Weeks) | 239; 13 teams | 198; 15 teams
Follow-Up #1 (6 Months) | 213; 13 teams | 163; 15 teams
Follow-Up #2 (12 Months) | 212; 13 teams | 174; 15 teams
Completed | 200; 13 teams | 152; 15 teams
Not Completed | 63; 0 teams | 66; 0 teams
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Injury | 2 | 0
Not completed — Kicked off team | 5 | 0
Not completed — Lost to Follow-up | 50 | 62

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Weight Intervention | Brochure Wait List | Total
Number analyzed (Participants) | 263 | 218 | 481
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.29 (1.25) | 19.42 (1.18) | 19.35 (1.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263 | 218 | 481
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 27 | 64
  Not Hispanic or Latino | 205 | 183 | 388
  Unknown or Not Reported | 21 | 8 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 7 | 2 | 9
  Native Hawaiian or Other Pacific Islander | 3 | 3 | 6
  Black or African American | 43 | 28 | 71
  White | 193 | 171 | 364
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 11 | 26
Height (inches) [Mean (Standard Deviation); unit: inches] | 65.95 (3.39) | 66.18 (4.00) | 66.05 (3.68)
Weight (pounds) [Mean (Standard Deviation); unit: pounds] — Self-reported
  pounds | 140.80 (22.47) | 138.80 (23.72) | 139.90 (23.04)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.74 (3.01) | 22.23 (2.65) | 22.50 (2.86)

OUTCOME MEASURES:

1. Primary Outcome: Eating Disorder Examination Questionnaire (EDE-Q)
Description: The Eating Disorder Examination Questionnaire (EDE-Q) assesses eating disorder behaviors through a self-report questionnaire. There are four subscales of the EDE-Q--Restraint, Eating Concern, Shape Concern, and Weight Concern--with scores for each ranging from 0-6. Overall scores also range from 0-6. Higher scores reflect greater severity of eating disorder psychopathology. Subscales are averaged to compute a total score.
Time Frame: 18 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Healthy Weight Intervention | Brochure Wait List
Number analyzed (Participants) | 263 | 218
units on a scale
  Global | .98 (.17) | 1.24 (.16)
  Restraint | .54 (.11) | .84 (.18)
  Shape Concern | 1.13 (.21) | 1.46 (.28)
  Weight Concern | 1.03 (.26) | 1.17 (.24)
  Eating Concern | .49 (.16) | .55 (.15)

2. Secondary Outcome: Secondary Outcomes
Description: Internalization of the Sport-Specific Thin-Ideal (ISTI) measures thin-ideal internalization specific to athletes (average of items from 1-5; higher scores mean worse outcome).
  Teammate Relationship Health (TRH) measures relational health with teammates (scores from 8-40; higher scores mean better outcome).
  Ideal-Body Stereotype Scale - Revised (IBSS-R) assesses internalization of the traditional thin-ideal (scores from 1-10, higher scores mean worse outcome).
  Positive and Negative Affect Scale - Revised (PANAS-X) assesses negative affect (average of items from 1-5; higher scores mean worse outcome).
  Intervention Suitability Expectations (ISE) assesses perceived suitability and expectations of the intervention (average of total scores from 4-46; higher scores mean better outcome).
  Knowledge of the Female Athlete Triad (KFAT) measures participant understanding of the Female Athlete Triad (each correct answer = 1, scores from 0-10; higher scores mean better outcome).
Time Frame: 18 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Healthy Weight Intervention | Brochure Wait List
Number analyzed (Participants) | 263 | 218
score on a scale
  Internalization of the Sport-Specific Thin-Ideal | 2.46 (.18) | 2.71 (.31)
  Teammate Relationship Health (TRH) | 30.28 (.65) | 29.87 (.85)
  Ideal-Body Stereotype Scale - Revised (IBSSR) | 3.20 (.06) | 3.43 (.05)
  Positive and Negative Affect Scale - Revised | 1.50 (.04) | 1.59 (.06)
  Intervention Suitability Expectations (ISE) | 29.92 (7.80) | 26.50 (8.52)
  Knowledge of the Female Athlete Triad | 8.54 (.37) | 8.58 (.30)

3. Primary Outcome: Number of Subjective and Objective Binge Episodes as Measured by the Eating Disorder Examination Questionnaire (EDE-Q)
Description: Frequency of subjective and objective binge episodes is reported.
Time Frame: 18 months
Measure: Mean (Standard Error); unit: episodes
Arm/Group | Healthy Weight Intervention | Brochure Wait List
Number analyzed (Participants) | 263 | 218
episodes
  Objective Binge Episode Frequency | .35 (1.56) | .63 (1.75)
  Subjective Binge Episode Frequency | .49 (1.94) | .57 (3.52)

4. Secondary Outcome: Secondary Outcomes - BMI
Description: Body Mass Index (BMI) (self-reported) is a measure of kg/m^2.
Time Frame: 18 months
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Healthy Weight Intervention | Brochure Wait List
Number analyzed (Participants) | 263 | 218
kg/m^2 | 25.09 (1.12) | 24.22 (.90)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a period of 18 months.
Description: Because this study involved the evaluation of an athlete prevention program via assessment measures, with oversight by the school athletic department, minimal risk was anticipated in this remote study. Adverse events related to the study (questionnaires) were monitored. Participants were also monitored by the school athletic department based on their previously established protocols.
Arm/Group | Healthy Weight Intervention | Brochure Wait List
All-Cause Mortality (participants affected / at risk) | 0/263 | 0/218
Serious Adverse Events (participants affected / at risk) | 0/263 | 0/218
Other Adverse Events (participants affected / at risk) | 0/263 | 0/218

LIMITATIONS AND CAVEATS:
The cluster randomized control trial design by team reduced statistical power. We could not control for team-based variability. Selective attrition may have occurred by the intervention of school athletic medical staff.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2013-07-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT01735994/Prot_000.pdf
  • Informed Consent Form (2013-07-10): https://cdn.clinicaltrials.gov/large-docs/94/NCT01735994/ICF_001.pdf
  • Statistical Analysis Plan (2019-09-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT01735994/SAP_002.pdf